CLINICAL TRIAL: NCT04231513
Title: A Randomized, Double-Blind, Placebo-Controlled, Combined Single Ascending Dose and Multiple Ascending Dose Study to Assess Safety, Tolerability, Pharmacokinetics, Immunogenicity, and Pharmacodynamics of Intravenous Infusions of E2814 in Healthy Subjects
Brief Title: A Study to Assess Safety, Tolerability, Pharmacokinetics (PK), Immunogenicity, and Pharmacodynamics (PD) of Intravenous Infusions of E2814 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Other
Other Study IDs: E2814-A001-001
Record Dates: First submitted 2020-01-14; First posted 2020-01-18 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Healthy Volunteers
Keywords: E2814; Healthy Participants; Phase 1; Pharmacokinetics; Pharmacodynamics; Immunogenicity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- SAD, Cohort 1: E2814 or E2814-matched Placebo (Experimental): Participants will receive either E2814 or E2814-matched placebo as an intravenous infusion, once, on Day 1.
  Interventions: Drug: E2814; Drug: E2814-matched placebo
- SAD, Cohort 2: E2814 or E2814-matched Placebo (Experimental): Participants will receive either E2814 or E2814-matched placebo as an intravenous infusion, once, on Day 1.
  Interventions: Drug: E2814; Drug: E2814-matched placebo
- SAD, Cohort 3: E2814 or E2814-matched Placebo (Experimental): Participants will receive either E2814 or E2814-matched placebo as an intravenous infusion, once, on Day 1.
  Interventions: Drug: E2814; Drug: E2814-matched placebo
- SAD, Cohort 4: E2814 or E2814-matched Placebo (Experimental): Participants will receive either E2814 or E2814-matched placebo as an intravenous infusion, once, on Day 1.
  Interventions: Drug: E2814; Drug: E2814-matched placebo
- SAD, Cohort 5: E2814 or E2814-matched Placebo (Experimental): Participants will receive either E2814 or E2814-matched placebo as an intravenous infusion, once, on Day 1.
  Interventions: Drug: E2814; Drug: E2814-matched placebo
- MAD, Cohort 1: E2814 or E2814-matched Placebo (Experimental): Participants will receive E2814 or E2814-matched placebo as an intravenous infusion Q4W on 3 occasions up to Day 57 of the Treatment Period.
  Interventions: Drug: E2814; Drug: E2814-matched placebo
- MAD, Cohort 2: E2814 or E2814-matched Placebo (Experimental): Participants will receive E2814 or E2814-matched placebo as an intravenous infusion Q4W on 3 occasions up to Day 57 of the Treatment Period.
  Interventions: Drug: E2814; Drug: E2814-matched placebo
- MAD, Cohort 3: E2814 or E2814-matched Placebo (Experimental): Participants will receive E2814 or E2814-matched placebo as an intravenous infusion Q4W on 3 occasions up to Day 57 of the Treatment Period.
  Interventions: Drug: E2814; Drug: E2814-matched placebo
- MAD, Cohort 4: E2814 or E2814-matched Placebo (Experimental): Participants will receive E2814 or E2814-matched placebo as an intravenous infusion Q4W on 3 occasions up to Day 57 of the Treatment Period.
  Interventions: Drug: E2814; Drug: E2814-matched placebo

INTERVENTIONS:
Drug: E2814 — E2814, intravenous infusion.
Drug: E2814-matched placebo — E2814-matched placebo, intravenous infusion.

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of single and multiple intravenous infusions of E2814 in healthy adult participants.

DETAILED DESCRIPTION:
The study is comprised of two components: a single ascending dose (SAD) component and a multiple ascending dose (MAD) component. The SAD component consists of 5 sequential cohorts and in each cohort, 8 healthy participants are randomized (3:1) to receive a single dose of E2814 or E2814-matched placebo. The MAD component of the study consists of 4 sequential cohorts and in each cohort, 8 healthy participants are randomized (3:1) to receive E2814 or E2814-matched placebo every 4 weeks (Q4W) on 3 occasions.

ELIGIBILITY:
Inclusion Criteria:

1. Nonsmoking, healthy participants.

Japanese participants must satisfy the following requirements:

1. Must have been born in Japan to Japanese parents and Japanese grandparents
2. Must have lived no more than 5 years outside of Japan
3. Must not have changed their life style or habits, including diet, while living outside of Japan

Exclusion Criteria:

1. Clinically significant illness that requires medical treatment within 8 weeks or a clinically significant infection that requires medical treatment within 4 weeks of dosing
2. Females who are breastfeeding or pregnant at Screening or Baseline
3. Females of childbearing potential who within 28 days before study entry, did not use a highly effective method of contraception, which includes any of the following:

   1. total abstinence (if it is their preferred and usual lifestyle)
   2. an intrauterine device or intrauterine hormone-releasing system
   3. a contraceptive implant
   4. an oral contraceptive (Participants must be on a stable dose of the same oral contraceptive product for at least 28 days before dosing and throughout the study and for 16 weeks after study drug discontinuation)
   5. have a vasectomized partner with confirmed azoospermia Do not agree to use a highly effective method of contraception (as described above) throughout the entire study period and for 16 weeks after study drug discontinuation NOTE: All females will be considered to be of childbearing potential unless they are postmenopausal (amenorrheic for at least 12 consecutive months, in the appropriate age group, and without other known or suspected cause) or have been sterilized surgically (that is, bilateral tubal ligation, total hysterectomy, or bilateral oophorectomy, all with surgery at least 1 month before dosing).
4. Males who have not had a successful vasectomy (confirmed azoospermia) or they and their female partners do not meet the criteria above (that is, not of childbearing potential or practicing highly effective contraception throughout the study period and for 5 times the half-life of the study drug plus 90 days after study drug discontinuation). If the female partner is pregnant, then males who do not agree to use latex, or synthetic condoms throughout the study period and for 90 days after study drug discontinuation. No sperm donation is allowed during the study period and for 5 times the half-life of the study drug plus 90 days after study drug discontinuation
5. Evidence of disease that may influence the outcome of the study within 4 weeks before dosing; example, psychiatric disorders and disorders of the gastrointestinal tract, liver, kidney, respiratory system, endocrine system, hematological system, neurological system, or cardiovascular system, or participants who have a congenital abnormality in metabolism
6. Any clinically abnormal symptom or organ impairment found by medical history, physical examinations, vital signs, ECG finding, or laboratory test results that requires medical treatment at Screening or Baseline
7. A prolonged QT (that is, corrected QT interval [QTc] Fridericia interval greater than [>] 450 milliseconds) demonstrated on ECG at Screening or Baseline. A history of risk factors for torsade de pointes (example, heart failure, hypokalemia, family history of long QT Syndrome)
8. Persistent systolic blood pressure (SBP) >130 millimeters of mercury (mmHg) or diastolic blood pressure (DBP) >85 mmHg at Screening or Baseline. One repeat measurement will be allowed
9. Heart rate less than 45 or more than 100 beats per minute at Screening or Baseline
10. Known history of clinically significant drug allergy at Screening or Baseline
11. Known history of food allergies or presently experiencing significant seasonal or perennial allergy at Screening or Baseline
12. Any history of hypersensitivity reaction to a foreign protein, with clinical features of Grades 2 to 4 as described in National Cancer Institute-Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0, immunoglobulin A (IgA) deficiency, or significant autoimmune disease or disorder. Participants with hypersensitivity reactions to foreign protein with clinical features limited to nasal or conjunctival symptoms such as in allergic rhinitis do not need to be excluded
13. Known to be human immunodeficiency virus (HIV) positive at Screening
14. Active or chronic (including asymptomatic) viral hepatitis (A, B or C) as demonstrated by positive serology at Screening. For hepatitis B serology, this refers to positive for hepatitis B core antibody (HBcAb, Immunoglobulin M [IgM] type) or hepatitis B surface or core antigens (HBsAg, HBcAg). For hepatitis C serology, a positive result for screening serological testing must be confirmed by qualitative hepatitis C virus ribonucleic acid (RNA)
15. History of drug or alcohol dependency or abuse within the 2 years before Screening, or those who have a positive urine drug test or breath (or urine) alcohol test at Screening or Baseline
16. Intake of over-the-counter medications within 2 weeks before dosing
17. Currently enrolled in another clinical study or used any investigational drug or device within 30 days (or 5 half-lives, whichever is longer) preceding informed consent
18. Exposure to any biologic drug within 90 days or at least 5 half-lives (whichever is longer), or within 4 weeks for vaccines, before Screening, with the exception of influenza and COVID-19 vaccinations that are allowed up to 7 days before dosing
19. Engagement in strenuous exercise within 2 weeks before check-in (example, marathon runners, weight lifters, etc.)
20. Any contraindication to continuous cerebrospinal fluid (CSF) sampling via indwelling lumbar catheter or via lumbar puncture (LP)
21. Any history of or current blood clotting or bleeding disorder that is not under adequate control, including a platelet count less than (<) 50,000, international normalized ratio (INR) >1.3, or partial thromboplastin time (PTT) >upper limit of normal (ULN), or fibrinogen <1.8 gram per liter (g/L) or >4.3 g/L at Screening or Baseline. Participants receiving anticoagulation therapy or identified at risk for hemorrhage
22. Any lifetime suicidal behavior or psychiatric disease. Whenever possible, medical records should be reviewed to confirm absence of history of psychiatric disease or use of medications to treat psychiatric disease
23. Any current or prior history of suicidal behavior or psychiatric disease identified by the psychiatrist at the Screening Visit

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2019-12-16 (Actual); Primary Completion 2023-03-09 (Actual); Study Completion 2023-03-09 (Actual)

PRIMARY OUTCOMES:
SAD, Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | Up to 113 days
SAD, Number of Participants With Clinically Significant Laboratory Values | Up to 113 days
SAD, Number of Participants With Clinically Significant Vital Signs Values | Up to 113 days
SAD, Number of Participants With Clinically Significant Electrocardiogram (ECG) Findings | Up to 113 days
MAD, Number of Participants With TEAEs and SAEs | Up to 169 days
MAD, Number of Participants With Clinically Significant Laboratory Values | Up to 169 days
MAD, Number of Participants With Clinically Significant Vital Signs Values | Up to 169 days
MAD, Number of Participants With Clinically Significant ECG Findings | Up to 169 days

SECONDARY OUTCOMES:
SAD, Cmax Serum: Maximum Observed Concentration for E2814 | Pre-dose (Day 1) and up to Day 113 Post Dose
SAD, Tmax Serum: Time to Reach the Maximum Observed Concentration (Cmax) for E2814 | Pre-dose (Day 1) and up to Day 113 Post Dose
SAD, AUC (0-24h) Serum: Area Under the Concentration-time Curve From Time Zero to 24 Hour for E2814 | Pre-dose (Day 1) and up to 24 hours Post Dose
SAD, AUC (0-72h) Serum: Area Under the Concentration-time Curve From Time Zero to 72 Hour for E2814 | Pre-dose (Day 1) and up to 72 hours Post Dose
SAD, AUC (0-inf) Serum: Area Under the Concentration-time Curve from Time 0 to Infinity for E2814 | Pre-dose (Day 1) and up to Day 113 Post Dose
SAD, t½ Serum: Terminal Elimination Phase Half-life for E2814 | Pre-dose (Day 1) and up to Day 113 Post Dose
SAD, CL Serum: Clearance for E2814 | Pre-dose (Day 1) and up to Day 113 Post Dose
SAD, Vz Serum: Volume of Distribution for E2814 | Pre-dose (Day 1) and up to Day 113 Post Dose
SAD, Serum anti-E2814 Antibody Concentration | Pre-dose (Day 1) and up to Day 113 Post Dose
SAD, Cmax CSF: Maximum Observed Concentration for E2814 | Pre-dose (Day 1) and up to Day 29 Post Dose
SAD, Tmax CSF: Time to Reach the Maximum Observed Concentration (Cmax) for E2814 | Pre-dose (Day 1) and up to Day 29 Post Dose
SAD, AUC (0-24h) CSF: Area Under the Concentration-time Curve From Time Zero to 24 Hour for E2814 | Pre-dose (Day 1) and up to 24 hours Post Dose
SAD, Cmax Plasma: Maximum Observed Concentration for E2814 | Pre-dose (Day 1) and up to Day 113 Post Dose
SAD, Tmax Plasma: Time to Reach the Maximum Observed Concentration (Cmax) for E2814 | Pre-dose (Day 1) and up to Day 113 Post Dose
SAD, AUC (0-24h) Plasma: Area Under the Concentration-time Curve From Time Zero to 24 Hour for E2814 | Pre-dose (Day 1) and up to 24 hours Post Dose
SAD, AUC (0-72h) Plasma: Area Under the Concentration-time Curve From Time Zero to 72 Hour for E2814 | Pre-dose (Day 1) and up to 72 hours Post Dose
SAD, AUC (0-inf) Plasma: Area Under the Concentration-time Curve from Time 0 to Infinity for E2814 | Pre-dose (Day 1) and up to Day 113 Post Dose
SAD, t½ Plasma: Terminal Elimination Phase Half-life for E2814 | Pre-dose (Day 1) and up to Day 113 Post Dose
SAD, CL Plasma: Clearance for E2814 | Pre-dose (Day 1) and up to Day 113 Post Dose
SAD, Vz Plasma: Volume of Distribution for E2814 | Pre-dose (Day 1) and up to Day 113 Post Dose
SAD, Plasma anti-E2814 Antibody Concentration | Pre-dose (Day 1) and up to Day 113 Post Dose
MAD, Cmax Serum: Maximum Observed Concentration for E2814 | Pre-dose (Day 1) and up to Day 169 Post Dose
MAD, Tmax Serum: Time to Reach the Maximum Observed Concentration (Cmax) for E2814 | Pre-dose (Day 1) and up to Day 169 Post Dose
MAD, AUC (0-24h) Serum: Area Under the Concentration-time Curve From Time Zero to 24 Hour for E2814 | Pre-dose (Day 1) and up to 24 hours Post Dose
MAD, AUC (0-72h) Serum: Area Under the Concentration-time Curve From Time Zero to 72 Hour for E2814 | Pre-dose (Day 1) and up to 72 hours Post Dose
MAD, AUC (0-tau) Serum: Area Under the Concentration-time Curve From Zero Time to the end of the Dosing Interval for E2814 | Pre-dose (Day 1) and up to Day 169 Post Dose
MAD, t½ Serum: Terminal Elimination Half-life for E2814 | Pre-dose (Day 1) and up to Day 169 Post Dose
MAD, CL Serum: Clearance for E2814 | Pre-dose (Day 1) and up to Day 169 Post Dose
MAD, Vz Serum: Volume of Distribution for E2814 | Pre-dose (Day 1) and up to Day 169 Post Dose
MAD, Rac(Cmax) Serum: Ratio of Accumulation for Cmax for E2814 | Pre-dose (Day 1) and up to Day 169 Post Dose
MAD, Rac(AUC) Serum: Ratio of Accumulation for AUC for E2814 | Pre-dose (Day 1) and up to Day 169 Post Dose
MAD, Serum anti-E2814 Antibody Concentration | Pre-dose (Day 1) and up to Day 169 Post Dose
MAD, CSF Concentration for E2814 | Pre-dose (Day 1) and up to Day 85 Post Dose
MAD, Cmax Plasma: Maximum Observed Concentration for E2814 | Pre-dose (Day 1) and up to Day 169 Post Dose
MAD, Tmax Plasma: Time to Reach the Maximum Observed Concentration (Cmax) for E2814 | Pre-dose (Day 1) and up to Day 169 Post Dose
MAD, AUC (0-24h) Plasma: Area Under the Concentration-time Curve From Time Zero to 24 Hour for E2814 | Pre-dose (Day 1) and up to 24 hours Post Dose
MAD, AUC (0-72h) Plasma: Area Under the Concentration-time Curve From Time Zero to 72 Hour for E2814 | Pre-dose (Day 1) and up to 72 hours Post Dose
MAD, AUC (0-tau) Plasma: Area Under the Concentration-time Curve From Zero Time to the end of the Dosing Interval for E2814 | Pre-dose (Day 1) and up to Day 169 Post Dose
MAD, t½ Plasma: Terminal Elimination Half-life for E2814 | Pre-dose (Day 1) and up to Day 169 Post Dose
MAD, CL Plasma: Clearance for E2814 | Pre-dose (Day 1) and up to Day 169 Post Dose
MAD, Vz Plasma: Volume of Distribution for E2814 | Pre-dose (Day 1) and up to Day 169 Post Dose
MAD, Rac(Cmax) Plasma: Ratio of Accumulation for Cmax for E2814 | Pre-dose (Day 1) and up to Day 169 Post Dose
MAD, Rac(AUC) Plasma: Ratio of Accumulation for AUC for E2814 | Pre-dose (Day 1) and up to Day 169 Post Dose
MAD, Plasma anti-E2814 Antibody Concentration | Pre-dose (Day 1) and up to Day 169 Post Dose

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - California Clinical Trials Medical Group/Parexel International, Glendale, California
  - Worldwide Clinical Trials, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.